CLINICAL TRIAL: NCT05055297
Title: SELUTION SLR™ 014 BTK: A Prospective Randomized Multicenter Single Blinded Study to Assess the Safety and Effectiveness of the SELUTION SLR™ 014 Drug Eluting Balloon in the Treatment of Below-the-Knee (BTK) Atherosclerotic Disease in Patients With Chronic Limb Threatening Ischemia (CLTI)
Brief Title: SELUTION4BTK Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.A. Med Alliance S.A. (Industry)
Collaborators: NAMSA (Other); Cordis US Corp. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: S2021-01
Record Dates: First submitted 2021-09-14; First posted 2021-09-24 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2025-11

CONDITIONS: Peripheral Arterial Disease; Chronic Limb-Threatening Ischemia Nos of Native Arteries of Extremities
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Angioplasty, Balloon

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- SELUTION SLR™ DEB 014 (Experimental)
  Interventions: Device: SELUTION SLR™ DEB 014
- Plain (Uncoated) Balloon Angioplasty (PTA) (Active Comparator)
  Interventions: Device: Plain (Uncoated) Balloon Angioplasty (PTA)

INTERVENTIONS:
Device: SELUTION SLR™ DEB 014 — a non-surgical procedure that uses a catheter to inflate a drug-eluting balloon to open up peripheral below-the-knee arteries that have been narrowed by chronic limb-threatening ischemia
  Arms: SELUTION SLR™ DEB 014
Device: Plain (Uncoated) Balloon Angioplasty (PTA) — a non-surgical procedure that uses a catheter to inflate a commercially available, non-drug-eluting balloon to open up peripheral below-the-knee arteries that have been narrowed by chronic limb-threatening ischemia
  Arms: Plain (Uncoated) Balloon Angioplasty (PTA)

SUMMARY:
This study aims to demonstrate superior efficacy and equivalent safety of the SELUTION SLR™ DEB 014 compared to plain (uncoated) balloon angioplasty in the treatment of peripheral arterial disease (PAD) in the BTK arteries in CLTI patients.

ELIGIBILITY:
Clinical Inclusion Criteria:

1. Subject age is ≥ 18 years or older depending on local regulations.
2. Subject life expectancy is ≥ 1 year.
3. Subject has documented chronic limb-threatening ischemia in the target limb with Rutherford classification category 4 or 5 and symptoms of > 2 weeks duration.
4. Subject is willing and able to provide written informed consent and comply with study procedures and required follow-up evaluations.
5. Female subjects of childbearing potential must be non-breastfeeding and have a negative pregnancy test ≤ 7 days before the procedure.

Angiographic Inclusion Criteria:

Subjects must meet all the following criteria to be enrolled in the trial:

1. Target lesion(s) must be de novo or non-stented restenotic lesion(s) located within the BTK arteries distal to the tibial plateau and above the tibiotalar joint line. BTK arteries include the P3 segment of the popliteal artery, the tibio-peroneal trunk, peroneal artery, anterior tibial artery, and posterior tibial artery.
2. BTK Target lesions cannot be contiguous with inflow lesions and at least 3 cm of normal artery should extend beyond the tibial plateau to ensure there is no overlap.
3. Target lesions must have a diameter stenosis of ≥ 70% (including total occlusions) by visual estimate and must be indicated for PTA treatment.
4. Target vessel reference diameter(s) are ≥ 2mm and ≤ 4mm. Note: the SELUTION SLR 014 DEB and the control PTA balloon size cannot exceed 4.0 mm.
5. Target lesions must be confined to a single target vessel. NOTE: Subjects with other non-target BTK lesions in separate non-target vessels may be enrolled, provided that the non-target lesions have been successfully treated (residual stenosis ≤ 30% with no distal embolization or flow limiting ≥ Grade C dissection). NOTE: Any adjunctive therapies are permitted for the treatment of non-target BTK lesions, but no DEB or DES may be used.
6. Any target lesion must be ≥ 30 mm in length and the total combined length of all target lesions must be ≤ 140 mm (total treatment length ≤ 150 mm allowing for 5 mm proximal and distal shoulder treatment). Note: All target lesions and all inflow lesions must be treatable by one or more SELUTION SLR 014/018 DEB(s) such that the total planned per-subject drug dose (calculated by summing the drug dose of all individual planned balloon sizes) would be ≤ 7069 μg. Note: A total treated segment length of ≤ 150 mm for BTK and ≤ 200 mm for inflow segment is acceptable irrespective of DEB balloon diameter.
7. The tibial and pedal runoff distal to the target lesions must be patent OR the target vessel(s) must reconstitute above the ankle or display normal terminal branching as follows:

   1. If the target vessel is the P3 segment, any 1 of the 3 distal arteries must show a patent (≤ 50% stenosis by visual estimate) outflow.
   2. If the target vessel is the peroneal artery, the artery must demonstrate normal terminal branching.
   3. If the target vessel is the anterior tibial (AT) or posterior tibial (PT) artery, the artery must reconstitute ≥ 1 cm above the tibiotalar joint to provide an intact runoff vessel (AT: dorsalis pedis; PT: plantar artery).
   4. If the target vessel is the tibio-peroneal trunk, outflow for either the peroneal OR the posterior tibial artery must be patent (≤ 50% stenosis by visual estimate).
8. Subjects is free of significant inflow vessel disease or any inflow disease has been successfully treated (see angiographic inclusion # 9). Significant inflow disease is defined as ≥ 50% stenosis by visual estimate. Inflow vessels include the ipsilateral common iliac, external iliac, common femoral, profunda femoris, superficial femoral or popliteal artery proximal (≥ 3 cm) to the tibial plateau. Note: If access site doesn't permit angiographic imaging of the common iliac and common femoral artery (CFA), then non-invasive imaging (CTA or MRA) must be provided to exclude presence of significant inflow disease. If non-invasive imaging is not possible, a DUS of the CFA with a multiphasic wave form excluding significant disease AND a palpable ipsilateral femoral pulse must be documented.
9. Subjects with significant inflow disease (≥ 50% stenosis by visual estimate) must have documented successful treatment before randomizing the subject. Successful treatment of inflow disease is defined as ≤ 30% final residual stenosis and no distal embolization or flow-limiting > Grade C dissection. Note: Treatment of the common femoral and profunda femoris is not permitted. Inflow vessel treatment can be performed with any commercially available non-DCB or non-DES device; if DCB treatment is required, SELUTION SLR 018 must be used.
10. The BTK target lesion preparation must be documented to be successful by angiography (≤ 30% residual stenosis and no distal embolization or flow-limiting ≥ Grade C dissection) before randomization. Note: Lesion preparation can include atherectomy (rotational, orbital, directional or laser), cutting, scoring, contoured balloons or intravascular lithotripsy and PTA only.

Clinical Exclusion Criteria:

Subjects will be excluded if any of the following criteria apply:

1. Subject has extensive tissue loss (Rutherford category 6) extending above the trans metatarsal level, salvageable only with complex foot reconstruction or non-traditional trans metatarsal amputations. This includes subjects with:

   1. Osteomyelitis involving proximal to the metatarsal head(s)
   2. Any heel wound or wound with calcaneal bone involvement

   d) Wounds that would require flap coverage or complex wound management for large soft tissue defect e) Full-thickness wounds on the dorsum of the foot with exposed tendon or bone
2. Subject has chronic renal insufficiency (dialysis dependent, or glomerular filtration rate [GFR] ≤ 30 ml/min/1.73 m2 within 30 days of index procedure) or has undergone renal transplantation.
3. Subject has acute renal insufficiency confirmed by 50% increase of serum creatinine within 48 hours before procedure and/or decrease in urine output.
4. Subject has acute limb ischemia with onset of index limb symptoms less than 2 weeks prior to index procedure.
5. Subjects has wounds that are deemed to be neuropathic or non-ischemic in nature or any venous or mixed wounds.
6. Subject has had prior major amputation of the ipsilateral extremity or planned major amputation of either leg.
7. Target limb iliac or common femoral artery bypass within 6 weeks of index procedure.
8. Prior (within 14 days) or planned (within 30 days) surgical or endovascular procedures. The following procedures are permitted:

   1. Target limb inflow treatment at the index procedure, provided it meets the criteria in Angiographic Inclusion Criteria #12
   2. Contralateral limb iliac artery treatment
   3. Diagnostic angiography
   4. Foot wound debridement
   5. Planned minor amputation of digit(s) at the phalangeal level
9. Target lesion has undergone prior DCB within 1 year, or ANY prior DES or bare metal stent (BMS) treatment (no in-stent restenosis [ISR] treatment is permitted). Note: Prior stent is permitted if the target lesion is located ≥ 30 mm from the stent AND there is ≤ 30% in-stent diameter stenosis.
10. Target lesion(s) requires treatment with alternative therapies such as thrombolysis, thrombus aspiration, stenting, cryoplasty, brachytherapy, or re-entry device. Note: The following adjunctive lesion preparation therapies are permitted: Atherectomy (rotational, orbital, directional or laser), cutting/scoring/contoured balloon, or intravascular lithotripsy.
11. Target lesion requires treatment via pedal access or upper extremity access.
12. Subject has undergone non-coronary artery treatment with any limus-based drug coated balloon (DCB) or DES or other device within 3 months prior to index procedure.
13. Subject has known hypersensitivity or allergy to Sirolimus or other pharmacologic agents required for the procedure (such as contrast agent, heparin, bivalirudin) that cannot be adequately pre-treated.
14. Subject has contraindication to antiplatelet therapy.
15. Subject has experienced disabling stroke or ST-segment elevation myocardial infarction (STEMI) within 3 months of index procedure.
16. Subject has acute coronary syndrome. Stabilized Acute Coronary Syndrome (ACS) is permitted.
17. Subject has non-atherosclerotic disease of the target vessel (including aneurysmal disease and vasculitis) or Buerger's disease.
18. Subject has hypercoagulable state or disorder, or coagulopathy, including platelet count ≤ 100,000 per microliter.
19. Subject has systemic infection (White Blood Count [WBC] > 12,000 and febrile). [Note: Enrollment permitted after successful treatment of infection with resolution of leukocytosis and/or febrile state].
20. Subject is known to be immune compromised (e.g., Human Immunodeficiency virus [HIV], Systemic Lupus Erythematosus [SLE]) or is receiving treatment with immune suppressive medications (NOTE: topical corticosteroids are permitted)
21. Subject is receiving (or is scheduled to receive) cancer treatment with surgery or chemotherapy or radiation therapy or has metastatic malignancy. Note: local application of chemotherapeutic creams is allowed.
22. Subject has New York Heart Association (NYHA) class IV congestive heart failure.
23. Subject is bedridden.
24. Subject has a body mass index (BMI) < 18.
25. Subject is currently participating in another investigational drug or device study that has not completed primary endpoint follow-up.
26. Subject has other anatomic, medical, social, or psychological conditions that in the investigator's opinion could limit the patient's ability to participate in the clinical study and/or comply with the follow-up requirements.

Angiographic Exclusion Criteria:

Subjects will be excluded if any of the following criteria apply:

1. Presence of a previously placed stent in the target vessel(s), UNLESS the target lesion is located ≥ 30 mm from the stent AND there is ≤ 30% in-stent diameter stenosis.
2. There is significant (> 50% diameter stenosis) inflow disease in the common femoral and profunda femoris arteries (inflow treatment of the common femoral and profunda femoris is not permitted).
3. The target lesion could not be successfully pre-dilated (residual stenosis > 30%, distal embolization, or flow-limiting ≥ Grade C dissection after pre-dilatation).
4. Intra-arterial thrombus, thromboembolism or atheroembolism in the index limb noted on initial diagnostic angiography or following treatment of inflow disease or pre-treatment of target lesion.
5. Subject requires treatment of the tibial arteries distal to the tibiotalar joint line, or treatment of the pedal arteries. Angioplasty at or below the tibiotalar joint is not permitted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 376 (Estimated)
Dates: Start 2022-05-19 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2032-07-30 (Estimated)

PRIMARY OUTCOMES:
Primary Efficacy Endpoint | 6 months
  Hierarchical composite efficacy endpoint determined by pair-wise comparisons among all subjects (Win Ratio method) according to the following pre-specified hierarchy of adverse outcomes:
  * Major (above-the-ankle) amputation
  * CD-TLR
  * Target lesion occlusion by angiography (if angiography is not available, the decision will be made on a secondary modality, in order of preference: computed tomography angiogram [CTA], magnetic resonance angiography [MRA] or DUS)
  * Transverse View Area Loss (TVAL%) by angiography.
Primary Safety Endpoint | 30 days
  Freedom from the composite of MALE and all-cause perioperative death (POD). MALE is defined as major (above-the-ankle) amputation or major reintervention (new bypass graft, jump/ interposition graft revision, thrombectomy/thrombolysis) of the index limb.

SECONDARY OUTCOMES:
Primary sustained clinical improvement | 1, 6, 12, 24, and 36 months
  A secondary efficacy endpoint defined as freedom from target limb major amputation and CD-TLR AND increase in Rutherford category from baseline.
Secondary sustained clinical improvement | 1, 6, 12, 24, and 36 months
  A secondary efficacy endpoint defined as freedom from target limb major amputation AND increase in Rutherford category from baseline.
Major amputation | 1, 6, 12, 24, and 36 months
  A secondary efficacy endpoint defined as above-the-ankle amputation of the target limb.
Amputation-free survival | 1, 6, 12, 24, and 36 months
  A secondary efficacy endpoint defined as freedom from all-cause mortality and major amputation.
Primary assisted patency | 1, 6, 12, 24, and 36 months
  A secondary efficacy endpoint defined as freedom from ACL adjudicated occlusion on angiography or, if angiography is not available, by CTA, MRA or Duplex ultrasound core laboratory (DCL) adjudicated duplex ultrasound, irrespective of interventions for stenoses.
  • Secondary patency, defined as freedom from permanent occlusion (occlusion at the last follow-up imaging) as determined by the ACL or DCL.
Secondary patency | 1, 6, 12, 24, and 36 months
  A secondary efficacy endpoint defined as freedom from permanent occlusion (occlusion at the last follow-up imaging) as determined by the ACL or DCL.
CD-TLR | 1, 6, 12, 24, and 36 months
  A secondary efficacy endpoint defined as re-intervention on target lesion(s) due to recurrent/persistent/worsening symptoms and the angiographic finding of ≥ 50% restenosis of target lesion by ACL measurement.
Clinically driven (CD-TVR) | 1, 6, 12, 24, and 36 months
  A secondary efficacy endpoint defined as re-intervention on target vessel due to recurrent/persistent/worsening symptoms and the angiographic finding of ≥ 50% restenosis of target vessel by ACL measurement.
Rutherford category | 1, 6, 12, 24, and 36 months
  A secondary efficacy endpoint defined as change in Rutherford category from baseline.
ABI/TBI/Toe Pressure | 1, 6, 12, 24, and 36 months
  A secondary efficacy endpoint defined as change in ankle brachial index (ABI), toe brachial index (TBI), and toe pressures from baseline.
  • Change in Quality of Life (QOL) measures from baseline (EQ-5D and VascuQol instruments)
Quality of Life (QOL) measures | 1, 6, 12, 24, and 36 months
  A secondary efficacy endpoint defined as change in Quality of Life (QOL) measures from baseline (EQ-5D and VascuQol instruments).
MALE | 1, 6, 12, 24, and 36 months
  A secondary safety endpoint defined as the composite of major (above-the-ankle) amputation or major reintervention (new bypass graft, jump/ interposition graft revision, thrombectomy/thrombolysis) of the index limb.
Major cardiovascular events | 1, 6, 12, 24, and 36 months
  A secondary safety endpoint defined as the composite of cardiovascular death, myocardial infarction (MI), and stroke.
  • All-cause mortality [evaluated at discharge, 1, 6, and 12 months and 2-5 years]
All-cause mortality | 1, 6, 12, 24, and 36 months
Device success | Post-procedure
  A secondary performance endpoint defined as successful delivery, balloon inflation, deflation and retrieval of the intact investigational device.
Procedural (technical) success | Post-procedure
  A secondary performance endpoint defined as device success and residual diameter stenosis ≤ 30% on completion angiography by core lab assessment.
Clinical success | Evaluated at discharge defined as immediately prior to hospital discharge from the index procedure or within 7 days, whichever occurs first
  A secondary performance endpoint defined as procedural success without procedural complications (death, above-ankle target limb amputation, thrombosis of the target lesion or TLR) prior to discharge.
Secondary Angiographic Imaging Measures | 6 months
  * Subsegmental analysis: proportion of segments with binary restenosis (DS > 50%)
  * Subsegmental analysis: Mean LLL of all segments; mean %DS of all segments.
  * TVAL%
Wound healing | 1, 6, 12, 24, and 36 months
  A secondary wound measure defined as investigator reported status of each index wound in comparison to baseline.
  Descriptive categories to be captured on case report forms (CRFs): 1) Improved 2) Unchanged 3) Worse 4) Healed/Complete Closure. Note: New wounds (appearing at any time after index procedure) are identified and tracked in similar fashion as index wounds, adopting the initial evaluation & images as "baseline" for future comparisons.
Wound Ischemia, foot infection (WifI) Classification | 1, 6, 12, 24, and 36 months
  A secondary wound measure defined as investigator-reported granular descriptors of Wound, Ischemia, and Foot Infection.

CONTACTS AND LOCATIONS:
Locations (48):
- United States (30):
  - Chandler Regional Medical Center, Chandler, Arizona
  - St. Bernards Medical Center, Jonesboro, Arkansas
  - Arkansas Heart Hospital, Little Rock, Arkansas
  - St. Helena Hospital, St. Helena, California
  - Lundquist Institute for Biomedical Innovation at Harbor UCLA Medical Center, Torrance, California
  - ClinRé, Thornton, Colorado
  - Vascular Care Group, Darien, Connecticut
  - Yale University, New Haven, Connecticut
  - The Cardiac and Vascular Institute Research Foundation, Gainesville, Florida
  - Palm Vascular Centers, Miami, Florida
  - Guardian Research Organization, LLC, Winter Park, Florida
  - Cardiovascular Consultants of South Georgia, Thomasville, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Cardiovascular Institute of the South, Gray, Louisiana
  - MedStar Health Research Institute, Hyattsville, Maryland
  - Beth Israel Medical Center, Boston, Massachusetts
  - University of Massachusetts Medical Center, Worcester, Massachusetts
  - Sorin Medical Group, New York, New York
  - NC Heart and Vascular Research, LLC, Raleigh, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Hightower Clinical Research, Oklahoma City, Oklahoma
  - Miriam Hospital, Providence, Rhode Island
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Tennessee Center for Clinical Trials, Tullahoma, Tennessee
  - El Paso Cardiology, El Paso, Texas
  - Baylor College of Medicine, Houston, Texas
  - Texas Cardiac and Vascular Institute San Antonio, San Antonio, Texas
  - Christus Health, Tyler, Texas
- LKH-Universitätsklinikum Graz, Graz, Austria
- France (2):
  - Ambroise Paré Hospital, Boulogne-Billancourt
  - Hôpital St. Joseph, Paris
- Germany (6):
  - Alexianer Klinikum Hochsauerland, Arnsberg
  - Universitäts-Herzzentrum Freiburg - Bad Krozingen, Bad Krozingen
  - Krankenhaus Buchholz, Buchholz
  - Sana Kliniken Oberfranken Coburg, Coburg
  - University of Essen, Essen
  - Universitatsklinikum Tubingen, Tübingen
- Hong Kong (2):
  - Queen Mary Hospital, Hong Kong, Pok Fu Lam
  - The Chinese University of Hong Kong, Hong Kong, Shatin
- Italy (3):
  - Ospedale Pederzoli, Peschiera del Garda, Verona
  - UGC - Maria Cecilia Hospital, Cotignola
  - Ospedale Policlinico San Martino, Genova
- St. Antonius Hospital, Nieuwegein, Netherlands
- Auckland City Hospital, Auckland, New Zealand
- Singapore General Hospital, Singapore, Singapore
- Inselspital Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No